CLINICAL TRIAL: NCT05453032
Title: Effects of Transcranial Direct Current Stimulation in Conjugation With Psychotherapy on Impulsivity in Patients With Borderline Personality Disorder
Brief Title: The Effect of Non Invasive Brain Stimulation on Impulsivity in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Dr. Lionel Cailhol, chef of psychiatry department at Montreal Psychiatric Institute (IUSMM) (Unknown)
Responsible Party: Principal Investigator, Ahmad Al Zatam, Master's Student, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2308
Record Dates: First submitted 2022-03-29; First posted 2022-07-12 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Borderline Personality Disorder
Keywords: impulsivity; Non-Invasive Brain Stimulation; Psychotherapy
MeSH Terms: conditions — Borderline Personality Disorder; Impulsive Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: we recruited 10 patients who attended a 10-session of tDCS stimulation. Each session lasted for 20 minutes in a 2-week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with BPD assigned to the trial of 10 active tDCS sessions followed by psychotherapy (Experimental): Patients diagnosed with Borderline Personality disorder and BPDSI score is > or = 17 will be assigned for active tDCS session (NeuroConn, Germany) candidates will have 20-minute session per day for 10 weekdays in 2 weeks. Then they will attend short term psychotherapy session for 3 months.
  Interventions: Device: NeuroConn

INTERVENTIONS:
Device: NeuroConn — A neurostimulation decivse that works be generating weak electric current via Electrodes. These electrodes placed on a specific cerebral location, where the defect assumed to be there) to modulate the neuronal activity. This neuronal modulation does not induce or fire action potential but it facilitate action potentials and cerebral interconnection as well corticolimbic connection)
  Other Names: tDCS; transcranial Direct Current Stimulation

SUMMARY:
A pilot study to examine the effects of Non-Invasive Brain stimulation on impulsive behaviour in patients diagnosed with Borderline Personality Disorder. patients who received the neurostimulation sessions will be enrolled in short term psychotherapy (3-month)

ELIGIBILITY:
Inclusion Criteria

* Clinical Diagnosis of Borderline Personality Disorder (DSM-V)
* Resident of Great Montreal
* Ability to make decision
* Clinical score is equal or more than 17 in Borderline Personality Disorder Severity Index (BPDSI)

resident of greater Montreal Area,

Exclusion Criteria:

* material Metal in the brain
* History of seizure or epilepsy
* severe scalp irritation or eczema
* recent scares, cut wounds, tattoo on the scalp
* severe substance use disorder
* clinical diagnosis of severe mood disorders o
* Active psychotic episode
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
The effect of NIBS on impulsivity (UPPS- Behavioral Impulsive scale) | 2-week stimulation session
  Patients with BPD will complete UPPS impulsive behavioral scale, a self reported questionnaire, before the first tDCS session and after they complete the 10 sessions of tDCS sessions. this questionnaire consists of 45 questions with 4 likert scale range for each question. The questionnaire is divided into 4 subscales: Urgency, lack of premeditation, lack of perseverance, sensation seeking.

SECONDARY OUTCOMES:
The effect of tDCS on BPD severity overall ( Borderline Personality Disorder Severity Index: BPDSI) | 3 months
  The BPD patients who attend the tDCS sessions and the short-term psychotherapy will be evaluated by one psychiatric with a semi-structured interview evaluation, Borderline Personality disorder Severity Index (BPDSI)
The Effect of tDCS on Risk taking ( an impulsive behavior dimension) | 2 weeks
  a computerized measure of risk taking behavior. Each participant will have a set of 30 balloons with temporary and permanent bank. The possibility of balloon explosion increased each time the participant inflate ( click on the balloon) while the amount of money increased by 0.5 euro with each inflation. the participant could more the earned money from inflation anytime before unexpected balloon explosion to the permanent bank. The total number of the pumps will determine the probability of risk taking behavior
the effect of tDCS on depressive symptoms in BPD (Montgomery-Asberg Depression Rating Scale (MADRS)) | 2 weeks
  A self reported questionnaire that assess the depressive symptoms in the last 3 days. it consists of 9 questions with 3 likert score range ; each question examines different aspect of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Recherche_ Institut Univesitaire de Santé Mentale à Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share the results only while keeping the coincidentally for the participants

REFERENCES:
- [Background] Lisoni J, Miotto P, Barlati S, Calza S, Crescini A, Deste G, Sacchetti E, Vita A. Change in core symptoms of borderline personality disorder by tDCS: A pilot study. Psychiatry Res. 2020 Sep;291:113261. doi: 10.1016/j.psychres.2020.113261. Epub 2020 Jun 28. PMID 32622171
- [Background] Lisoni J, Barlati S, Deste G, Ceraso A, Nibbio G, Baldacci G, Vita A. Efficacy and tolerability of Brain Stimulation interventions in Borderline Personality Disorder: state of the art and future perspectives - A systematic review. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Jun 8;116:110537. doi: 10.1016/j.pnpbp.2022.110537. Epub 2022 Feb 15. PMID 35176417
- [Result] Teti Mayer J, Chopard G, Nicolier M, Gabriel D, Masse C, Giustiniani J, Vandel P, Haffen E, Bennabi D. Can transcranial direct current stimulation (tDCS) improve impulsivity in healthy and psychiatric adult populations? A systematic review. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Mar 2;98:109814. doi: 10.1016/j.pnpbp.2019.109814. Epub 2019 Nov 9. PMID 31715284